CLINICAL TRIAL: NCT01476982
Title: Evaluation of Patients in Chest Pain in the Emergency Room
Acronym: EPIC-ER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Epic Research & Diagnostics, Inc. (Industry)
Collaborators: Scottsdale Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC-001
Record Dates: First submitted 2011-10-28; First posted 2011-11-22 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Acute Cardiac Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Emergency Department Patients: Patients presenting to the Emergency Department complaining of chest pain.
  Interventions: Device: ClearView Scan

INTERVENTIONS:
Device: ClearView Scan — Assessment with ClearView device

SUMMARY:
The primary objective of this feasibility study is to determine whether it is possible to conduct a study of the ClearView scan among patients under evaluation for acute cardiovascular events, as well as give insight into the performance of the ClearView scoring algorithm with respect to this patient population. The EPIC™ scan is a bio-electrographic tool that may assist the health care provider in rapid assessment of the systemic origin of the patient's presenting symptom(s). The EPIC ClearView is a potentially valuable resource that may benefit an emergency department (ED) by offering expedited "chest pain" etiologic differentiation capabilities. The subsequent results have the potential to include more rapid "chest pain" patient diagnosis and appropriate disposition of non-cardiac chest pain (rule out MI); optimized precious resource expenditure (nursing, physician, inpatient or observation bed, etc.); lower costs to facility, patient and insurance company; and greater patient satisfaction rates due to decreased ED wait time.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: Male or Female
2. Age range: 18 to 85
3. Chief complaint upon admission to the ED: chest pain
4. The patient or legal representative is able to understand and provide signed consent for the procedure.
5. Every effort will be given to balance subjects by gender, age, and race.

Exclusion Criteria:

1. Patients < 18 years in age or > 85 years in age.
2. Inability or unwillingness to provide informed consent.
3. Patients with pacemakers or another electrical device, such as an automatic internal cardiac defibrillator, implanted somewhere in their body.
4. Patients connected to an electrical device that cannot be removed (i.e. monitor).
5. Pregnant women.
6. Patients currently undergoing therapy for cancer of any kind.
7. Patients missing all or part of any of their fingers.
8. Patients with hand tremors or involuntary oscillations ("shaking") of the hands that prevent clear imaging.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women, ages 18-85, presenting to the Emergency Department with chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Agreement of ClearView scan versus Active (Presenting) Diagnosis | At time of study scan (Single study visit only, with no follow-up. The study endpoint will be reported for day 0, the day of the study visit.)
  Statistical agreement will be assessed between the 0-25 ClearView Response Scale and the presenting diagnosis/diagnoses for the Emergency Department admission recorded within the medical record, on a per-subject basis.

CONTACTS AND LOCATIONS:
Overall Officials: Krishnaswami Vijayaraghavan, MD, Principal Investigator — Scottsdale Healthcare
Locations (2):
- United States (2):
  - Scottsdale Healthcare Osborn Campus, Scottsdale, Arizona
  - Scottsdale Healthcare Shea Campus, Scottsdale, Arizona